CLINICAL TRIAL: NCT03195387
Title: A Single Site, Randomized, Double-blind, Placebo-controlled Phase Ib Study, to Evaluate the Chemoprotective Activity of a Single Dose of MMV390048 in a Controlled P. Falciparum Sporozoite Infection Model in Non-immune Healthy Volunteers
Brief Title: Chemoprotective Activity of MMV390048 in PfSPZ Challenge Model
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Repositioning of target indication.
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Datamap (Industry); PrimeVigilance Zagreb (Unknown); ICON Clinical Research (Industry); Sanaria Inc. (Industry); PTx Solutions Ltd., UK (Unknown); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMV_MMV390048_17_01; 2017-002034-23 (EudraCT Number)
Record Dates: First submitted 2017-06-15; First posted 2017-06-22 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Malaria,Falciparum
Keywords: malaria, P. falciparum, chemoprotection, Phase Ib
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — MMV390048

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- D-1/120 mg MMV390048 (Experimental): Treatment of cohort 1: subjects receive a single oral dose of MMV390048 on Day -1, prior to PfSPZ challenge on Day 0.
  Interventions: Drug: MMV390048
- D-7/120 mg MMV390048 (Experimental): Treatment of cohort 2: subjects receive a single oral dose of MMV390048 on Day -7, prior to PfSPZ challenge on Day 0.
  Interventions: Drug: MMV390048
- D-X/YY mg MMV390048 (Experimental): Treatment of cohort 3: subjects receive a single oral dose of MMV390048 (dose to be determined) on a day (to be determined) prior to PfSPZ challenge on Day 0. Dosage and day of administration will be determined on the basis of data emerging from the first two cohorts.
  Interventions: Drug: MMV390048
- Placebo (Placebo Comparator): MMV390048 placebo
  Interventions: Drug: MMV390048

INTERVENTIONS:
Drug: MMV390048 — Each tablet contains 20 mg MMV390048 and the following excipients: tartaric acid powder, copovidone (Plasdone S-630), hypromellose acetate succinate (AquaSolve HPMC-AS MF), croscaramellose sodium (Solutab), microcrystalline cellulose type 102 (Avicel PH-102), magnesium stearate (Ligamed MF-2-V).
  Other Names: MMV-048

SUMMARY:
This study follows a First-In-Human dose-escalation study of MMV390048 (5 to 120 mg MMV390048 powder-in-bottle formulation), a formulation bioavailability study to establish suitable tablet formulation, and a two-part dose-escalation (40 to 120 mg of MMV390048) / induced blood stage malaria (ISBM) challenge study with the new tablet formulation. After identification of the predicted efficacious MMV390048 plasma concentrations in the IBSM model, the current study will evaluate the chemoprotective efficacy of MMV390048 in a standardised and validated controlled human malaria infection (CHMI) model using direct venous inoculation (DVI) of aseptic, purified, cryopreserved, vialed P. falciparum sporozoites (PfSPZ Challenge).

Three sequential cohorts of healthy men and women of non-childbearing potential (WONCBP) will be administered the investigational medicinal product (IMP, i.e. MMV390048) under different conditions. This may identify preventative regimens, to be further investigated in a Phase II program. In the first two cohorts, protective administration of the IMP will occur 1 and 7 days before DVI of PfSPZ challenge. The timing of IMP administration and dosage in the last cohort will be determined on the basis of emerging data from the preceding cohorts, but will not exceed 28 days prior to the challenge nor 120 mg MMV390048.

DETAILED DESCRIPTION:
Subjects are enrolled into one of three cohorts of 12 subjects each. Cohorts are recruited sequentially, to facilitate on-going review of data.

Investigational medicinal product (IMP) administration takes place between 28 and 1 days before the P. falciparum sporozoites (PfSPZ) challenge. Subjects are randomised to receive either MMV390048 120 mg or placebo in a 3:1 ratio.

After IMP administration, each subject is inoculated with 3200 PfSPZ. The dose of IMP to be administered and the interval between IMP administration and the PfSPZ challenge are as follows:

* Cohort 1: Subjects receive a single oral dose of MMV390048 (9 subjects) or placebo (3 subjects) on Day -1, prior to PfSPZ challenge on Day 0.
* Cohort 2: Subjects receive a single oral dose of MMV390048 (9 subjects) or placebo (3 subjects) on Day -7, prior to PfSPZ Challenge on Day 0.
* Cohort 3: Subjects receive a single oral dose of MMV390048 (9 subjects; dose to be determined) or placebo (3 subjects) on a day (to be determined) prior to PfSPZ challenge on Day 0. IMP dosage and day of administration will be determined on the basis of data emerging from the first two cohorts, but will not exceed 120 mg nor 28 days prior to PfSPZ challenge.

Parasitaemia and malaria symptoms and signs are monitored daily from Day 6 and as long as subjects exhibit parasitaemia (defined as either a positive thick blood smear microscopy or three positive quantitative polymerase chain reactions at least 12 hours apart with one measurement greater 100 parasites per mL), or until Day 28 if no parasitemia is not detected. All subjects receive antimalarial rescue therapy upon positive parasitaemia or at the end of the treatment period if parasites are not detected during follow-up. A final safety follow-up visit takes place on Day 60.

After treating cohorts 1 and 2 (up to, and including Day 28 assessments), a safety review team (SRT) meeting takes place, to consider enrolment of the subsequent cohort. At the first meeting, the SRT reviews safety and parasitaemia data to Day 28 and determines whether progression to treatment of cohort 2 is indicated. If no safety concerns are identified by the SRT and the geometric mean time to parasitaemia is less than 12 days for Cohort 1, progression to Cohort 2 takes place. Should Cohort 2 be enrolled, safety and parasitaemia data to Day 28 and PK data to at least Day 14 from this cohort are reviewed by the SRT prior to enrolling Cohort 3.

Recruitment of cohort 3 will be put on hold if:

* Any inoculum- or MMV390048-related SAEs are reported, or
* Two or more MMV390048-related severe (Grade 3 or higher) adverse events are reported in the same organ class, or
* Any significant inoculum-related adverse event is reported which may place subjects in a subsequent cohort at risk, or
* Any other critical findings are identified which may place subjects in a subsequent cohort at risk.

Dosing of a subsequent cohort at the same or lower dose with the same or increased interval between dosing and inoculation, will not be performed if:

• The cohort-specific geometric mean time to parasitaemia is less than 12 days.

If progression of the study to recruiting cohort 3 is approved the by SRT, the optimal dose of MMV390048, as well as the time point of its administration will be estimated based on PK modelling, using data from all trials and assuming that asexual liver and blood stage have similar MMV390048 sensitivities.

ELIGIBILITY:
Inclusion Criteria:

* Completion of written informed consent for study participation by the volunteer
* Able and willing to answer all questions on the informed consent quiz correctly, demonstrating an understanding of the study information and of the procedures associated with the study
* Men or WONCBP aged ≥ 18 and ≤ 45 at screening
* Good health based on the absence of significant medical history and clinically significant findings on physical examination and special investigations at screening and prior to IMP administration
* Body mass index >18 and < 30 [kg/m2]
* Negative alcohol breath test and urine drug screening test at screening (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates) and upon admission prior to IMP administration
* Sexually active male volunteers with female partners must agree to use a highly effective, medically acceptable form of contraception from the day of IMP administration until 120 days thereafter (covering a full sperm cycle of 90 days starting after 5 x t½ of the drug). Abstinent male volunteers or male volunteers with same-sex partners must agree to use the above-mentioned contraceptive methods if they commence heterosexual relations during the study, and to continue these methods until 120 days after IMP administration. Acceptable methods of contraception include the following:

  * Condom and occlusive cap (diaphragm or cervical/vault caps)
  * Surgical sterilization (vasectomy with documentation of azoospermia) plus utilisation of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps])
  * The subject's female partner uses contraception known to inhibit ovulation (combined oral oestrogen/progesterone preparation, oral or injectable progesterone, subdermal implants or transdermal contraceptive patch) commenced at least 14 days prior to IMP administration to the male subject plus utilisation of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps]
  * The subject's female partner has undergone documented bilateral tubal ligation (female sterilization) plus utilisation of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps]
  * The subject's female partner has undergone documented placement of an intrauterine device or intrauterine system plus utilisation of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps]
* Women must be of non-childbearing potential as per one of the following definitions:

  * surgically sterile (by hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy) as documented by a surgical report or by ultrasound, or
  * post-menopausal (spontaneous amenorrhoea for ≥ 12 months, or spontaneous amenorrhoea for 6-12 months and follicle-stimulating hormone (FSH) ≥ 40 IU/mL; either should be together with the absence of oral contraceptive use for > 12 months)
* Consent to permit the investigators to discuss the volunteer's medical history with their General Practitioner and to sign a request to release medical information concerning contraindications for participation in the study
* Able and willing (in the investigator's opinion) to comply with all study requirements for the duration of the study
* Agreement to undergo all study procedures, to attend all study visits and stay overnight for observations as required, up to and including the last follow-up visit
* Willingness to undergo a CHMI by DVI with PfSPZ Challenge
* Reachable (24/7) by mobile phone or electronic mail during the whole study period
* Agreement to refrain from blood donation during the course of the study and after the end of their involvement in the study according to the local and national blood banking eligibility criteria (currently 4 years in Germany)
* Willingness to take a curative regimen of artemether-lumefantrine (Riamet®) or another registered antimalarial if necessary

Exclusion Criteria:

* Any history of malaria
* Volunteer has travelled to or lived in a malaria-endemic area for more than 4 weeks during the 12 months prior to IMP administration, or spent any time in an endemic area during the 4 weeks prior to IMP administration
* Plans to travel to malaria endemic region during the study period up to last follow-up visit
* Plans to travel outside of Germany during the challenge period
* Volunteer is unable to be closely followed for social, geographic or psychological reasons
* Previous participation in any malaria vaccine or CHMI study
* Previous participation in a trial with MMV390048
* Participation in any other clinical study within 30 days or five half-lives of the investigational compound in that study (whichever is longer) prior to IMP administration in this study, or plans to participate in other investigational vaccine/drug research during the study period
* Participation in any research study involving blood sampling during the 8 weeks prior to IMP administration. (Volunteers from whom blood was last drawn at least 4 weeks prior to IMP administration, and from whom less than 450 ml of blood was taken during the 8 weeks leading up to the last study-related blood draw, may be considered on a case by case basis by the Investigator.)
* Blood product donation to any blood bank during the 8 weeks (whole blood) or 4 weeks (plasma and platelets) prior to IMP administration
* Blood loss of more than 100 ml during the 4 weeks prior to IMP administration
* Male volunteers with a female partner(s) who is (are) pregnant or lactating at the time of the administration of the IMP
* Women of childbearing potential, or nursing (lactating) women
* Positive HIV, HBV (seropositive for hepatitis B surface antigen) or HCV tests
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection, asplenia (e.g. post-splenectomy), recurrent, severe infections, or the use of chronic (more than 14 days) immunosuppressant or immune-modifying drugs within the 6 months prior to IMP administration. (The use of oral antihistamines, topical steroids or inhaled steroids at doses less than the equivalent of 800 ug budesonide or 750 ug fluticasone daily are not classified as immunosuppressant or immune-modifying for the purpose of this criterion.)
* History of serious psychiatric condition that may affect participation in the study or preclude compliance with the protocol, including but not limited to past or present psychoses, disorders requiring lithium, a history of attempted or planned suicide, more than one previous episode of major depression, any previous single episode of major depression lasting for or requiring treatment for more than 6 months, or any episode of major depression during the 5 years preceding screening. The Beck Depression Inventory will be used as an objective tool for the assessment of depression at screening. In addition to the conditions listed above, subjects with a score of 20 or more on the Beck Depression Inventory and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. Subjects with a Beck score of 17 to 19 may be enrolled at the discretion of the Investigator if they do not have a history of the psychiatric conditions mentioned in this criterion and their mental state is not considered to pose additional risk to the health of the volunteer or to the execution of the study and interpretation of the data gathered
* History of convulsions or of severe head trauma
* History of frequent headaches (either severe in nature or requiring continuous daily treatment or treatment more than three times per week on average) and/or migraines
* A history of clinically significant systemic disorders including haematological, renal, endocrine, gastrointestinal, hepatic, cardiovascular, pulmonary, dermatological, neurological, immunological or other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* History of cancer (except localised basal cell carcinoma of the skin)
* History of diabetes mellitus
* History of asthma
* Falling in moderate or higher risk category for a fatal or non-fatal cardiovascular event within 5 years (> 10%) determined by non-invasive criteria for cardiac risk
* History of arrhythmias or documented prolonged QTcB- or QTcF-interval (> 450 msec), any previous episode of syncope thought to be of cardiac origin, or a family history of long QT syndrome or unexplained sudden death
* Positive family history of cardiac disease in first and second degree relatives < 50 years
* Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g. recurrent episodes of fainting, palpitations, etc.)
* Any surgical or medical condition possibly affecting drug absorption (e.g. cholecystectomy, gastrectomy, bowel disease), distribution, metabolism or excretion
* History or presence of diagnosed food or known drug allergies (including but not limited to allergy to any of the antimalarial rescue medications to be used in the study), or history of anaphylaxis or other severe allergic reactions. (Subjects with seasonal allergies that are untreated and asymptomatic at the time of dosing will not be excluded.)
* History of psoriasis or porphyria
* Sickle cell anaemia or other red blood cell disorders
* G6PD deficiency
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including haematological, renal, endocrine, gastrointestinal, hepatic, cardiovascular, pulmonary, dermatological, neurological, immunological or other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* Resting vital signs (measured after 5 minutes in the supine position) at screening, admission to the CCT, or baseline prior to IMP administration as follows:

  * Tympanic body temperature ≥ 38.0 °C
  * SBP ≤ 90 or ≥ 140 mmHg
  * DBP ≤ 50 or ≥ 90 mmHg
  * Pulse rate ≤ 40 or ≥ 100 bpm Vital signs measurement may be repeated once in assessing this criterion if the investigator believes that the values from the original measurement were erroneous
* Symptomatic postural hypotension at screening, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg 2 minutes after changing from a supine to standing position
* Clinically significant abnormalities in electrocardiogram at screening, admission to the CCT, or baseline prior to IMP administration as follows:

  * PR-interval >210 msec
  * QRS-complex >120 msec
  * QTcB- or QTcF-interval >450 msec
  * pathologic Q wave
  * significant ST-T wave changes
  * left or right ventricular hypertrophy
  * non-sinus rhythm except isolated premature atrial contractions
  * incomplete left bundle branch block, or complete or intermittent right or left bundle branch block
  * second or third degree A-V heart block The ECG reading may be repeated once in assessing this criterion if the investigator believes that the values from the original reading were erroneous.
* Haematology, clinical chemistry, coagulation or urinalysis results at screening or on admission to the CCT prior to IMP administration that are outside of Sponsor-approved clinically acceptable laboratory ranges documented prior to study start or are considered clinically relevant
* Contraindications to the use of chloroquine phosphate, atovaquone-proguanil, artemether or lumefantrine
* Use of any prescription drugs, herbal supplements (e.g. St John's Wort), or over-the-counter medication within 7 days or five half-lives (whichever is longer) prior to IMP administration, or an anticipated requirement for the use of these during the course of the study. (If necessary, the incidental use of NSAIDs, vitamins and topical treatments may be acceptable after approval by the study Sponsor and will be documented in the case report form [CRF]. The use of nutritional supplements during this time that are not believed to have the potential to affect subject safety nor the overall results of the study, may be permitted on a case-by-case basis following approval by the Sponsor in consultation with the Investigator.)
* Use of systemic antibiotics with known antimalarial activity within 30 days of IMP administration (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, or azithromycin) or an anticipated requirement for the use of these during the study period
* Use of medications known to interact with chloroquine, atovaquone-proguanil (Malarone®) or artemether-lumefatrine (Riamet®) such as cimetidine, metoclopramide or antacids, or an anticipated requirement for the use of these at any point during the study period
* Ingestion of any poppy seeds within 24 hours prior to the screening or pre-dose urine drug screen
* Intake of grapefruit or grapefruit juice within 5 days of IMP administration, or unwillingness to abstain from the consumption of these products from 5 days prior to IMP administration until collection of the final PK blood sample
* Use of immunoglobulins or blood products within 3 months prior to IMP administration
* Suspected or known history of, or current alcohol abuse, or heavy intake defined as greater than 28 g (men) or 18 g (women) per day or a carbohydrate deficient transferrin level ≥ 2.5%
* Current drug habituation, or suspected or known intravenous drug abuse in the 5 years preceding enrolment
* Current smoking of more than 10 cigarettes or equivalent per day and/or unwilling to abstain from smoking during the admission period
* Plan for major surgery between enrolment and completion of study follow-up
* Personnel (e.g. investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study
* The subject has been committed to an institution by virtue of an order issued by either the judicial or administrative authorities

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cohort-specific geometric mean time to parasitaemia | Up to 28 days
  Defined by a positive thick blood smear (with 2 qualified microscopists detecting 2 unambiguous parasites each) or qPCR (three positive measurements, each at least 12 hours apart and one with parasitaemia greater 100 parasites per mL), or Day 28 if there is no parasitaemia.

SECONDARY OUTCOMES:
Incidence, severity and relationship to MMV390048 of the observed and self-reported treatment-emergent adverse events | Until Day 29 after IMP administration (cohort-dependent)
  Safety and tolerability assessments during 29 days after administration of a single oral dose of IMP.
Malaria clinical score and incidence, severity and relationship of the observed and self-reported adverse events after PfSPZ challenge | From PfSPZ challenge to the day of positive parasitaemia and to Day 28 and Day 60 (EOS visit)
  Safety and tolerability of the PfSPZ challenge in non-immune healthy volunteers.
Area under the plasma concentration-time curve from time zero to time of last measurable concentration (AUClast) | Duration of the PK study is up to 29 days after IMP administration
  Estimation of PK parameters using non-compartmental methods after a single oral dose of MMV390048.
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | Duration of the PK study is up to 29 days after IMP administration
  Estimation of PK parameters using non-compartmental methods after a single oral dose of MMV390048.
Maximum plasma drug concentration (Cmax) | Duration of the PK study is up to 29 days after IMP administration
  Estimation of PK parameters using non-compartmental methods after a single oral dose of MMV390048.
Time to reach maximum plasma drug concentration following administration (Tmax) | Duration of the PK study is up to 29 days after IMP administration
  Estimation of PK parameters using non-compartmental methods after a single oral dose of MMV390048.
Elimination half-life (t1/2) | Duration of the PK study is up to 29 days after IMP administration
  Estimation of PK parameters using non-compartmental methods after a single oral dose of MMV390048.
Apparent total drug clearance from plasma after oral administration (CL/F) | Duration of the PK study is up to 29 days after IMP administration
  Estimation of PK parameters using non-compartmental methods after a single oral dose of MMV390048.
Apparent volume of distribution during terminal phase (Vz/F) | Duration of the PK study is up to 29 days after IMP administration
  Estimation of PK parameters using non-compartmental methods after a single oral dose of MMV390048.
MMV390048 plasma concentration upon PfSPZ challenge | One-off assessment
  Estimation of MMV390048 plasma concentration on the day of PfSPZ inoculation.
Time to installment of parasitaemia | Up to 28 days
  Characterisation of the relationship between MMV390048 exposure and time of installment of P. falciparum parasitaemia assessed by qPCR after PfSPZ challenge.

OTHER OUTCOMES:
Parasite multiplication rate during early asexual blood stage | Day 0 to day 60
  Estimation of the effect of MMV390048 on sporozoite multiplication rate by qPCR and statistical modelling.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Mordmüller, Dr, Principal Investigator — Institute of Tropical Medicine / Centre for Clinical Trials, Eberhard Karls University
Locations (1):
- Institute of Tropical Medicine / Centre for Clinical Trials, Eberhard Karls University, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sulyok M, Ruckle T, Roth A, Murbeth RE, Chalon S, Kerr N, Samec SS, Gobeau N, Calle CL, Ibanez J, Sulyok Z, Held J, Gebru T, Granados P, Bruckner S, Nguetse C, Mengue J, Lalremruata A, Sim BKL, Hoffman SL, Mohrle JJ, Kremsner PG, Mordmuller B. DSM265 for Plasmodium falciparum chemoprophylaxis: a randomised, double blinded, phase 1 trial with controlled human malaria infection. Lancet Infect Dis. 2017 Jun;17(6):636-644. doi: 10.1016/S1473-3099(17)30139-1. Epub 2017 Mar 28. PMID 28363637
- [Background] Mordmuller B, Supan C, Sim KL, Gomez-Perez GP, Ospina Salazar CL, Held J, Bolte S, Esen M, Tschan S, Joanny F, Lamsfus Calle C, Lohr SJ, Lalremruata A, Gunasekera A, James ER, Billingsley PF, Richman A, Chakravarty S, Legarda A, Munoz J, Antonijoan RM, Ballester MR, Hoffman SL, Alonso PL, Kremsner PG. Direct venous inoculation of Plasmodium falciparum sporozoites for controlled human malaria infection: a dose-finding trial in two centres. Malar J. 2015 Mar 18;14:117. doi: 10.1186/s12936-015-0628-0. PMID 25889522
- [Background] World Health Organization. World Malaria Report 2015. World Health. 2015;243